CLINICAL TRIAL: NCT04648176
Title: Evaluation of Surgical and Functional Results of the Application of MOSES Technology in the Holmium Laser Prostate Enucleation as a Treatment for Tract Symptoms Lower Urinary Secondary to Benign Prostatic Hyperplasia
Brief Title: Application of MOSES Technology in BPH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR(AG)501/2019
Record Dates: First submitted 2020-03-06; First posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Benign Prostatic Hyperplasia (BPH); Lower Urinary Tract Symptoms
Keywords: laser; Holmium; HoLEP; Moses
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HoLEP (Active Comparator): Conventional laser
  Interventions: Device: Moses technology
- m-HoLEP (Experimental): Moses technology
  Interventions: Device: Moses technology

INTERVENTIONS:
Device: Moses technology — Using Holmium laser with Moses technology or conventional one

SUMMARY:
In this study the investigators intend to compare the surgical and functional results of two different modalities of the use of the Holmium laser in prostate enucleation.

DETAILED DESCRIPTION:
In this study the investigators intend to compare the surgical and functional results of two different modalities of the use of the Holmium laser in prostate enucleation using MOSES technology.

ELIGIBILITY:
Inclusion Criteria:

* Prostatic volume between 70-200cc
* Acceptance to participate in the study.

Exclusion Criteria:

* Previous urethra stricture
* Previous prostate surgery
* Neurogenic bladder
* Bladder tumor
* Neurological disease with repercussion in the lower urinary tract.
* Severe psychiatric illness
* Inability of the patient to consent

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-03-06 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | 24 hours after the surgery
  Hemoglobin change

SECONDARY OUTCOMES:
Enucleation time | during the surgery
  Enucleation time change
Hemostasis time | during the surgery
  Hemostasis time change
Morcellating time | during the surgery
  Morcellating time change
Surgery time | during the surgery
  Surgery time change
Irrigated volume of serum | during the surgery
  Irrigated volume of serum change
complication rate | one month after the surgery
  difference of complication rate
urinary tract infection | one month after the surgery
  urinary tract infection rate differences
lower urinary tract symptoms | through study completion, an average of 3 years
  lower urinary tract symptoms rate differences
sexual function | through study completion, an average of 3 years
  sexual function differences

CONTACTS AND LOCATIONS:
Overall Officials: José Placer Santos, PhD, Principal Investigator — Vall d'Hebrón University Hospital
Locations (1):
- Vall d'Hebron University Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No